CLINICAL TRIAL: NCT04299503
Title: Phase 2 Double Blind Randomized Placebo Controlled Trial of Topical Crisaborole in Patients with Mild-to-Moderate Alopecia Areata
Brief Title: Topical Crisaborole in Patients with Alopecia Areata
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to identify subjects to meet inclusion criteria
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13289
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2022-01

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — crisaborole

STUDY DESIGN:
Intervention Model Description: Double-Blind Period: Weeks 0-12; Open-Label Period: Weeks 12-24
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All site staff will be masked with the exception of pharmacy staff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Crisaborole (Active Comparator): ointment applied topically in the morning and in the evening
  Interventions: Drug: Crisaborole Topical Ointment
- Placebo (Placebo Comparator): ointment applied topically in the morning and in the evening
  Interventions: Drug: Placebo Topical Ointment

INTERVENTIONS:
Drug: Crisaborole Topical Ointment — For every 10% of scalp affected, approximately ½ finger tip of study drug will be needed to cover the area with a thin layer. After the first application at baseline, the tubes will be weighed to determine the dose needed to cover the affected area. This will be the subject's target dose throughout the study
  Other Names: Eucrisa
  Arms: Crisaborole
Drug: Placebo Topical Ointment — For every 10% of scalp affected, approximately ½ finger tip of study drug will be needed to cover the area with a thin layer. After the first application at baseline, the tubes will be weighed to determine the dose needed to cover the affected area. This will be the subject's target dose throughout the study
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to determine whether topical crisaborole improves hair growth in alopecia areata.

DETAILED DESCRIPTION:
Each individual will be enrolled in the study for 24 weeks. Following a 28 days screening period, eligible subjects will be randomized in a 1:1 ratio to receive either crisaborole 2% ointment or matching placebo for 12 weeks. The primary endpoint is assessed at week 12. At the week 12 visit, all subjects will enter the open label treatment period where they will all receive crisaborole 2% ointment for an additional 12 weeks, with the last study visit taking place on week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent document indicating the subject has been informed of all aspects of the study.
2. Subject is willing and able to comply with scheduled visits, treatment plan, study drug administration, and other study procedures.
3. Clinical diagnosis of alopecia areata with at least one lesion 1 cm in diameter and no more than 20% of total scalp surface area.
4. Females of child-bearing potential agree to use a reliable method of birth control or remain absent during the study and for at least 4 weeks following the last dose of the assigned treatment.
5. If receiving concomitant medications for any reason, must be on a stable regimen and willing to stay on a stable regimen.
6. All treatments for alopecia areata are prohibited during the course of the study. If subjects received any of the following treatments, the minimum criteria are observed:

   * Must be discontinued for at least 12 weeks prior to Baseline:

     o Any investigational or experimental therapy or procedure for alopecia areata;
   * Exception: Investigational biologics should be discussed with Sponsor to confirm period of discontinuation required. Must be discontinued for at least 8 weeks prior to Baseline:

     o Laser or light based alopecia areata treatments
   * Must be discontinued for at least 4 weeks prior to Baseline:

     * Immunomodulating or immunosuppressive oral medications (corticosteroids, methotrexate, cyclosporine, etc.) Subjects who require these medications during the study (e.g. use of corticosteroids for a chronic obstructive pulmonary disease exacerbation) will be terminated from the study.
     * Injections of steroids to alopecia areata areas
     * Contact sensitization treatment
     * Oral minoxidil
     * Patients already taking finesteride for at least 3 months to treat conditions in addition to or other than hair loss (benign prostate hypertrophy, hormonal suppression, etc.) may continue on this medication so long as the dose remains stable throughout the study.
   * Must be discontinued for at least 2 weeks prior to Baseline:

     * Topical treatments that may affect alopecia areata, e.g., corticosteroids, topical tacrolimus/pimecrolimus, retinoids. Use of these medications in non-AA areas, for non-AA conditions is allowed.
     * Hair regrowth products containing minoxidil
   * Use of any prior and concomitant therapy not listed above which, in the opinion of the PI may interfere with the objective of the study, within 60 days prior to the Screening Visit is prohibited

Exclusion Criteria:

1. Other skin conditions that, in the opinion of the PI would interfere with evaluation of alopecia areata. Conditions may include other types of hair loss, including discoid lupus, lichen planus pilaris, frontal fibrosing alopecia, cicatricial alopecia, and trichotillomania (hair pulling).
2. Pregnant/breastfeeding females, or females of childbearing potential not using highly effective contraception. Women of childbearing potential must test negative for pregnancy and use contraception for at least four weeks after last dose of drug.
3. Current or recent history of clinically significant medical or psychiatric condition, which, in the judgment of the principal investigator, may increase risk associated with the study participation or drug administration. Examples include, but are not limited to, recent infections or injuries of the scalp.
4. Have a history of infection requiring parenteral or oral or topical antimicrobial therapy within 2 weeks prior to baseline.
5. Received a prohibited concomitant medication within 7 days or 5 half-lives (whichever is longer) prior to baseline visit.
6. Subjects who have had an allergic reaction (e.g. urticarial, anaphylactic) to crisaborole will be excluded.
7. Participated in a trial for a topical or oral JAK inhibitor. JAK inhibitors are thought to improve alopecia areata, and sometimes the effects of JAK inhibitors can last long after treatment is completed. Past treatment with these agents could confound the results of crisaborole's effectiveness for alopecia.
8. Is currently on an oral PDE4 inhibitor or oral JAK inhibitor. PDE4 inhibitors and JAK inhibitors have been theorized to improve alopecia. Treatment with these agents could confound our results on the effectiveness of crisaborole for alopecia areata.
9. Have participated in other research studies of investigational products within 4 weeks or 5 half-lives (whichever is longer) of the investigational product prior to baseline. Subjects cannot participate in studies of other investigational or experimental therapies or procedures at any time during their participation in this study.
10. Subjects who are investigational site staff members or relatives of those site staff members or subjects who are Sponsor employees directly involved in the conduct of the trial.
11. In the opinion of the investigator or Sponsor, the subject is inappropriate for entry into this study, or unwilling/unable to comply with study procedures and lifestyle guidelines.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Severity of Alopecia Tool (SALT) Score Double-Blind Period | Baseline to Week 12
  percent change in Severity of Alopecia Tool (SALT) score from baseline to Week 12. The range in score is 0% (no hair loss) to 100% (complete hair loss).
Severity of Alopecia Tool (SALT) Open-Label Period | Baseline to Week 24
  percent change in Severity of Alopecia Tool (SALT) score from baseline to Week 24. The range in score is 0% (no hair loss) to 100% (complete hair loss).

SECONDARY OUTCOMES:
Severity of Alopecia Tool (SALT)50 Response Double-Blind Period | Week 6 and Week 12
  Greater than or equal to 50% reduction in Severity of Alopecia Tool (SALT) score response in terminal hair at Week 6 and Week 12. The range in score is 0% (no hair loss) to 100% (complete hair loss).
Severity of Alopecia Tool (SALT)50 Response Open-Label Period | Week 24
  Greater than or equal to 50% reduction in Severity of Alopecia Tool (SALT) score response in terminal hair at Week 24. The range in score is 0% (no hair loss) to 100% (complete hair loss).
Severity of Alopecia Tool (SALT)90 Response Double-Blind Period | Week 6 and Week 12
  Greater than or equal to 90% reduction in Severity of Alopecia Tool (SALT) score response in terminal hair at Week 6 and Week 12. The range in score is 0% (no hair loss) to 100% (complete hair loss).
Severity of Alopecia Tool (SALT)90 Response Open-Label Period | Week 24
  Greater than or equal to 90% reduction in Severity of Alopecia Tool (SALT) score response in terminal hair at Week 24. The range in score is 0% (no hair loss) to 100% (complete hair loss).
alopecia areata Physician Global Assessment (aaPGA) Double-Blind Period | Week 6 and Week 12
  achieving an alopecia areata Physician Global Assessment (aaPGA) score of 3 or above at Weeks 6 and 12; (0 =no regrowth; 1 = <25% of regrowth; 2 = 25%-49% of regrowth; 3 = 50%-74% of regrowth; 4 = 75%-99% of re- growth; 5 = 100% of regrowth)
alopecia areata Physician Global Assessment (aaPGA) Open-Label Period | Week 24
  achieving an alopecia areata Physician Global Assessment (aaPGA) score of 3 or above at Week 24; (0 =no regrowth; 1 = <25% of regrowth; 2 = 25%-49% of regrowth; 3 = 50%-74% of regrowth; 4 = 75%-99% of re- growth; 5 = 100% of regrowth)
Alopecia Areata Symptom Impact Scale (AASIS) Double-Blind Period | Week 6 and Week 12
  percent change from Baseline in the Alopecia Areata Symptom Impact Scale (AASIS) at Week 6 and Week 12
Alopecia Areata Symptom Impact Scale (AASIS) Open-Label Period | Week 24
  percent change from Baseline in the Alopecia Areata Symptom Impact Scale (AASIS) at Week 24
Dermatology Life Quality Index (DLQI) Double-Blind Period | Week 6 and Week 12
  Percent change from Baseline in the Dermatology Life Quality Index (DLQI) at Week 6 and Week 12
Dermatology Life Quality Index (DLQI) Open-Label Period | Week 24
  Percent change from Baseline in the Dermatology Life Quality Index (DLQI) at Week 24

CONTACTS AND LOCATIONS:
Overall Officials: David Rosmarin, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Department of Dermatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No